CLINICAL TRIAL: NCT06965179
Title: The Impact of Game Activities on Life Satisfaction and Psychological Well-Being in Older Adults
Acronym: Game4elders
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, AYSUN KAZAK, PhD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 78017789/050.01.04/3072208
Record Dates: First submitted 2025-05-01; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Elderly; Game; Well Being
Keywords: Elderly; Jenga; Bocce game; life satisfaction; Psychological Well-Being
MeSH Terms: conditions — Personal Satisfaction; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study is planned to be conducted with a total of 36 volunteer participants, with 12 individuals in each group that meets the inclusion criteria (Jenga game group, Bocce game group, and control group)."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jenga game group (Experimental): In the Jenga game group, participants will complete the Elderly Information Form and Mini-Mental State Examination (MMSE) before the intervention. As pre-tests, the Life Satisfaction Scale (LSS) and the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) will also be administered. Participants will play Jenga in pairs for at least 30 minutes once a week over four weeks. Grouping will consider participant preferences and promote social interaction. After the intervention, the same scales (LSS and WEMWBS) will be re-administered as post-tests to evaluate changes in life satisfaction and mental well-being.
  Interventions: Other: Jenga game
- Bocce game group (Experimental): In the Bocce game group, participants will first complete the Elderly Information Form and Mini-Mental State Examination (MMSE), followed by pre-tests including the SF-36, Life Satisfaction Scale (LSS), and the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). Bocce sessions will take place once a week for four weeks, with each session lasting at least 30 minutes. Games will be played in pairs to enhance social interaction and psychomotor skills. Participants will be randomly assigned to six groups of two, considering individual preferences. Pairings will rotate weekly based on game outcomes to encourage diverse interaction. After the final week, the LSS and WEMWBS will be re-administered as post-tests by the researcher.
  Interventions: Other: Bocce game
- Control group (No Intervention): In the control group, participants will complete the Elderly Information Form and Mini-Mental State Examination (MMSE), along with pre-tests including the Life Satisfaction Scale (LSS) and the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). These participants will continue receiving the institution's standard care without any additional intervention from the researcher. At the end of the fourth week, the LSS and WEMWBS will be re-administered as post-tests.

INTERVENTIONS:
Other: Jenga game — In the Jenga game group, participants will complete the Elderly Information Form and Mini-Mental State Examination (MMSE) before the intervention. As pre-tests, the Life Satisfaction Scale (LSS) and the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) will also be administered. Participants will play Jenga in pairs for at least 30 minutes once a week over four weeks. Grouping will consider participant preferences and promote social interaction. After the intervention, the same scales (LSS and WEMWBS) will be re-administered as post-tests to evaluate changes in life satisfaction and mental well-being.
  Other Names: intervention group 1
  Arms: Jenga game group
Other: Bocce game — In the Bocce game group, participants will first complete the Elderly Information Form and Mini-Mental State Examination (MMSE), followed by pre-tests including the SF-36, Life Satisfaction Scale (LSS), and the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). Bocce sessions will take place once a week for four weeks, with each session lasting at least 30 minutes. Games will be played in pairs to enhance social interaction and psychomotor skills. Participants will be randomly assigned to six groups of two, considering individual preferences. Pairings will rotate weekly based on game outcomes to encourage diverse interaction. After the final week, the LSS and WEMWBS will be re-administered as post-tests by the researcher.
  Arms: Bocce game group

SUMMARY:
The rapid global increase in the elderly population has made supportive interventions for enhancing quality of life and psychological well-being in older adults increasingly important. Physical activity not only improves physiological functioning but also positively impacts mental health in the elderly. Exercise and even light physical activity contribute to reduced depressive symptoms, improved quality of life, and increased social engagement. Game-based activities such as bocce and Jenga encourage physical movement while also supporting cognitive functioning, thereby enhancing psychological well-being. Although relatively new in Türkiye, bocce has been utilized in nursing homes to promote active aging, while Jenga is a mentally stimulating activity known to improve cognitive performance. In this context, the impact of game-based interventions on life satisfaction and psychological well-being has gained significance. Nurses play a crucial role in facilitating older adults' participation in such activities, supporting their holistic care, and enhancing their well-being. The aim of this study is to investigate the effects of game-based activities-specifically bocce and Jenga-on life satisfaction, quality of life, and psychological well-being among older adults.

ELIGIBILITY:
Inclusion Criteria:

* Be 60 years old or older

Be literate

Not have visual or hearing impairments

Be able to communicate verbally

Not have sensory loss, arthritis, phlebitis, inflammation, eczema, fractures, etc.

Not have any loss of fingers or limbs

Have a score of 25 or higher on the Standardized Mini-Mental State Examination (SMMSE)

Not have been diagnosed with mental illnesses such as Parkinson's, Alzheimer's, or major depression

Be enrolled in the 60+ Lifelong University

Agree to participate in the study

Exclusion Criteria:Be 85 years old or older (35)

Have sensory problems in the hands

Have deformities in the hands and nails

Have open wounds or burns on the hands

Have limb loss in the fingers

Have neuropathy

-

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Psychological Well-Being | Pre-intervention and 5th week post-intervention
  The scale was developed by Tennant et al. (2007) to assess the mental well-being levels of the general population in the United Kingdom. It is a unidimensional, 14-item, 5-point Likert-type scale. Participants respond to each item using the following options: 1 = Strongly disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Strongly agree. The total score ranges from 14 to 70, with higher scores indicating higher levels of psychological well-being.
Life Satisfaction | Pre-intervention and 5th week post-intervention
  The "Satisfaction with Life Scale" (SWLS), developed by Diener, Emmons, Larsen, and Griffin (1985), consists of five items to assess individuals' life satisfaction. The scale is a Likert-type instrument, with responses ranging from "strongly disagree" to "strongly agree," and is scored on a 1-7 point scale. The total score can range from 5 to 35, with higher scores indicating higher life satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tse MMY, Lau JL, Kwan R, Cheung D, Tang ASK, Ng SSM, Lee PH, Yeung SSY. Effects of play activities program for nursing home residents with dementia on pain and psychological well-being: Cluster randomized controlled trial. Geriatr Gerontol Int. 2018 Oct;18(10):1485-1490. doi: 10.1111/ggi.13509. Epub 2018 Sep 25. PMID 30255637